CLINICAL TRIAL: NCT03588884
Title: An Open-Label, Repeated-Dose Safety, Efficacy, Pharmacokinetic and Pharmacodynamic Study of Oral CTAP101 Capsules, Immediate- Release (IR) Calcifediol, High-Dose Cholecalciferol, and Paricalcitol Plus Low-Dose Cholecalciferol in Patients With Secondary Hyperparathyroidism, Stage 3 or 4 Chronic Kidney Disease and Vitamin D Insufficiency
Brief Title: Repeated-dose Safety, Efficacy, Pharmacokinetic and Pharmacodynamic of CTAP101, Immediate-release Calcifediol, High-dose Cholecalciferol, and Paricalcitol Plus Low-dose Cholecalciferol in Patients With Secondary Hyperparathyroidism, Chronic Kidney Disease 3-4 and Vitamin D Insufficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTAP101-CL-4001
Record Dates: First submitted 2018-06-28; First posted 2018-07-17 (Actual); Results first posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Secondary Hyperparathyroidism Due to Renal Causes; Vitamin D Insufficiency; CKD Stage 3; CKD Stage 4
MeSH Terms: interventions — Calcifediol; Cholecalciferol; paricalcitol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CTAP101 (Active Comparator): CTAP101/Calcifediol Capsules 60 micrograms (mcg) once daily at bedtime, except on Days 1 and 29 when dosing will occur in the morning before breakfast
  Interventions: Drug: Calcifediol Oral Capsule
- Immediate-release (IR) calcifediol (Experimental): Immediate-release (IR) calcifediol/266 micrograms (mcg) capsule before breakfast on the mornings of Day 1 and Day 29
  Interventions: Drug: Calcifediol Oral Product
- Cholecalciferol (Experimental): Cholecalciferol/Capsules 300,000 International Units (IU) (high-dose) before breakfast on the mornings of Day 1 and Day 29
  Interventions: Drug: Cholecalciferol
- Paricalcitol (Active Comparator): Paricalcitol/Capsules 1 mcg plus cholecalciferol capsules 800 IU (low-dose) once daily in the morning before breakfast, except on Days 1 and29 when dosing will occur before breakfast
  Interventions: Drug: Cholecalciferol; Drug: Paricalcitol Oral Capsule

INTERVENTIONS:
Drug: Calcifediol Oral Capsule — Capsule, daily
  Other Names: CTAP101
  Arms: CTAP101
Drug: Calcifediol Oral Product — Capsule, once a month
  Arms: Immediate-release (IR) calcifediol
Drug: Cholecalciferol — Capsule, once a month
  Arms: Cholecalciferol; Paricalcitol
Drug: Paricalcitol Oral Capsule — Capsule, daily
  Arms: Paricalcitol

SUMMARY:
An Open-Label, Repeated-Dose Safety, Efficacy, Pharmacokinetic and Pharmacodynamic Study of Oral CTAP101 Capsules, Immediate- Release (IR) Calcifediol, High-Dose Cholecalciferol, and Paricalcitol Plus Low-Dose Cholecalciferol in Patients with Secondary Hyperparathyroidism, Stage 3 or 4 Chronic Kidney Disease and Vitamin D Insufficiency

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age.
2. Have stage 3 or 4 CKD (estimated glomerular filtration rate [eGFR] of ≥15 to <60 millilter per minute per 1.73 meter square (mL/min/1.73 m2) using the Modification of Diet in Renal Disease equation).
3. Be without any disease state or physical condition that might impair evaluation of safety and efficacy or which, in the Investigator's opinion, would interfere with study participation, including:

   1. Serum albumin ≤ 3.0 (grams per deciliter (g/dL);
   2. Serum transaminase (alanine transaminase, glutamic pyruvic transaminase, aspartate aminotransferase or glutamic oxaloacetic transaminase) > 2.5 times the upper limit of normal at screening; and,
   3. Urinary albumin excretion ≤3000 microgram per milligram (μg/mg) creatinine.
4. Exhibit during the initial screening visit:

   1. Plasma intact parathyroid hormone (iPTH) ≥70 picogram per milliliter (pg/mL) and <400 pg/mL if receiving calcitriol or other 1α- hydroxylated vitamin D analog (paricalcitol or doxercalciferol); or
   2. Plasma iPTH ≥100 pg/mL and <500 pg/mL if not receiving calcitriol or other 1α- hydroxylated vitamin D analog; and,
   3. Serum total 25-hydroxyvitamin D <30 nanogram per milliliter (ng/mL).
5. If taking calcitriol, other 1α-hydroxylated vitamin D analog, or vitamin D supplementation, must forgo treatment with these non-study agents for the duration of the study and undergo a 4-week washout period.
6. Exhibit after the 4-week washout period (if required):

   1. Plasma iPTH ≥100 pg/mL and <500 pg/mL;
   2. Corrected serum calcium <9.8 mg/dL; (corrected for serum albumin)
   3. Serum total 25-hydroxyvitamin D <30 nanogram per milliliter (ng/mL); and,
   4. Serum phosphorus <5.5 milligram per deciliter (mg/dL).
7. If taking more than 1,500 milligram per day (mg/day) of elemental calcium, reduce calcium use (to approximately 1,000 to ≤1,500 mg/day) for the duration of the study.
8. Willing and able to comply with study instructions and commit to all clinic visits for the duration of the study.
9. Female subjects of childbearing potential must be neither pregnant nor lactating and must have negative blood pregnancy tests at the first screening visit.
10. All female subjects of childbearing potential and male subjects with female partners of childbearing potential must agree to use effective contraception (implants, injectables, combined oral contraceptives, intrauterine device, sexual abstinence, vasectomy or vasectomized partner) for the duration of the study.
11. Be able to read, understand and sign the subject Informed Consent Form (ICF) or have a legal authorized representative (LAR) sign the ICF.

Exclusion Criteria:

1. History of or planned kidney transplant or parathyroidectomy
2. History (prior 3 months) of corrected serum calcium ≥9.8 mg/dL or serum phosphorus ≥5.5 mg/dL if not receiving calcitriol or other 1α-hydroxylated vitamin D analog.
3. Need for phosphate binders to maintain the serum phosphate < 5.5 mg/dL or use of phosphate binders within 4 weeks prior to screening
4. Use of calcimimetic therapy (cinacalcet or etelcalcetide) within 12 weeks of screening.
5. Receipt of bisphosphonate therapy or other bone modifying treatment within 6 months prior to enrollment.
6. Known previous or concomitant serious illness or medical condition, such as malignancy, human immunodeficiency virus, significant gastrointestinal or hepatic disease, intestinal malabsorption disorder, hepatitis or cardiovascular event that in the opinion of the Investigator may worsen or reduce life expectancy, and/or interfere with participation in the study.
7. History of neurological/psychiatric disorder, including psychotic disorder or dementia, or any reason which, in the opinion of the Investigator makes adherence to a treatment or follow-up schedule unlikely.
8. Known or suspected hypersensitivity to any of the constituents of the study drugs.
9. Currently participating in, or has participated in, an interventional/investigational study within 30 days prior to study screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - National Institute of Clinical Research, Inc., Garden Grove, California
  - Research by Design, LLC, Chicago, Illinois
  - Spaulding Clinical Research, West Bend, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CTAP101 | Immediate-release (IR) Calcifediol | Cholecalciferol | Paricalcitol
Started | 18 | 18 | 18 | 15
Completed | 18 | 15 | 15 | 14
Not Completed | 0 | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CTAP101 | Immediate-release (IR) Calcifediol | Cholecalciferol | Paricalcitol | Total
Number analyzed (Participants) | 18 | 18 | 18 | 15 | 69
Age, Continuous [Mean (Standard Deviation); unit: Year] | 67.1 (10.7) | 70.1 (14.4) | 67.9 (9.8) | 63.4 (12.0) | 67.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 5 | 10 | 32
  Male | 7 | 12 | 13 | 5 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 1 | 4
  Not Hispanic or Latino | 17 | 17 | 17 | 14 | 65
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Treatment-Emergent Adverse Events (TEAE) as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Description: This study is descriptive and no primary or secondary efficacy endpoints are defined.
Time Frame: 5 months
Measure: Number; unit: number of TEAE count
Arm/Group | CTAP101 | Immediate-release (IR) Calcifediol | Cholecalciferol | Paricalcitol
Number analyzed (Participants) | 18 | 18 | 18 | 15
number of TEAE count
  Grade 1 Mild | 39 | 12 | 13 | 10
  Grade 2 Moderate | 1 | 3 | 8 | 5
  Grade 3 Severe | 2 | 3 | 0 | 1
  Grade Potentially Life Threatening | 0 | 0 | 0 | 0
  Grade 5 Fatal | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | CTAP101 | Immediate-release (IR) Calcifediol | Cholecalciferol | Paricalcitol
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/18 | 2/18 | 4/18 | 1/15
Other Adverse Events (participants affected / at risk) | 7/18 | 7/18 | 8/18 | 8/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CTAP101 (N=18) | Immediate-release (IR) Calcifediol (N=18) | Cholecalciferol (N=18) | Paricalcitol (N=15)
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Quadrantanopia (Nervous system disorders) | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Blister (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CTAP101 (N=18) | Immediate-release (IR) Calcifediol (N=18) | Cholecalciferol (N=18) | Paricalcitol (N=15)
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Quadrantanopia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0
Tenderness (General disorders) | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Some institution and PI have the right to publish info 12 months after the study ended. For one PI that all Confidential Information must be held secret for a period of 5 years after end of the relevant Work Order.

DOCUMENTS (2):
  • Study Protocol (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT03588884/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT03588884/SAP_001.pdf